CLINICAL TRIAL: NCT01411748
Title: Comparison of Saccharomyces Boulardii and Nystatin Prophylaxis on Candida Colonization and Infection in Very Low Birth Weight Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Maternity and Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: demirel98
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-07

CONDITIONS: Anticandidal Property of Saccharomyces Boulardii on Very Low Birth Weight Infants

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S. boulardii (Experimental): The patients in this group will be given 5 million unit/day S. boulardii until discharge.
  Interventions: Dietary Supplement: Reflor
- nystatin (Active Comparator)
  Interventions: Drug: mikostatin

INTERVENTIONS:
Dietary Supplement: Reflor — 5 million unit/day, orally, beginning on the second day of life, until discharge from hospital
  Arms: S. boulardii
Drug: mikostatin — 50000 unit/3 times a day, both for orally and by orogastric route
  Arms: nystatin

SUMMARY:
Probiotics are favorable microorganisms that regulate the flora of the gastrointestinal system and stimulate the immune system. Saccharomyces boulardii was shown to reduce candida colonization. The objective of this study is to evaluate the efficacy of prophylactic S boulardii in reducing the candida colonization and infection in very low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants < 1500 gr

Exclusion Criteria:

* Genetic anomalies
* Not willing to participate
* Allergy to S. boulardii components

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of prophylactic S. boulardii and nystatin on candida colonization and infection in very low birth weight infants | 6 months

SECONDARY OUTCOMES:
Effect of S. boulardii on sepsis | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Division of Neonatology, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Chapman RL. Prevention and treatment of Candida infections in neonates. Semin Perinatol. 2007 Feb;31(1):39-46. doi: 10.1053/j.semperi.2007.01.006. PMID 17317426
- [Background] Murzyn A, Krasowska A, Stefanowicz P, Dziadkowiec D, Lukaszewicz M. Capric acid secreted by S. boulardii inhibits C. albicans filamentous growth, adhesion and biofilm formation. PLoS One. 2010 Aug 10;5(8):e12050. doi: 10.1371/journal.pone.0012050. PMID 20706577